CLINICAL TRIAL: NCT03888209
Title: Transcranial Direct Current Stimulation ASsociated With Physical-therapy In Acute Stroke Patients - the tDCS ASAP - a Randomized, Triple Blind, Sham-controlled Study ?
Brief Title: Transcranial Direct Current Stimulation (tDCS) Improves Functional Outcomes in Acute Stroke Patients
Acronym: tDCS ASAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-287
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Stroke, Acute
Keywords: tDCS; WMFT; Semmes Weinstein; Acute stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: randomized, triple blind, sham controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The device is preprogrammed by a third party non participating in any element in the study. They then chose (using opaque envelopes) the treatment code for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Experimental): Patients will receive 20min anodal tDCS
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Patients will receive 20 minutes of Sham anodal tDCS
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 20 minutes of anodal tDCS (C3/FP2 or C4/FP1 depending on side of lesion) 2mA or sham
  Other Names: Non invasive brain stimulation

SUMMARY:
Acute stroke patient will undergo one month (20 sessions) of physical therapy and anodal tDCS.

Patients will undergo functional outcomes measured at 48h post onset, 7,14,21,28 days, 3 and 6 months and one year post onset.

DETAILED DESCRIPTION:
Recruitment :

Patients with acute stroke (24-48h after stroke) who have upper and / or lower sensorimotor deficits

• Treatment : After being selected according to the inclusion and exclusion criteria of this study, patients will be randomized and placed in one of two groups: placebo (P) or transcranial anodic stimulation (A).

Once placed in one of two groups, patients will all receive intensive physiotherapy for functional improvement in order to increase motor, postural and motor control. This physiotherapy will be established 5 times a week (Monday to Friday).

In addition to physiotherapy, the patient will have electrodes placed on his head, attached via a system of straps, to deliver either a continuous current (A) or no current (P) and at a rate of 5 times per week for 4 weeks. Neither the physiotherapist nor the patient will know what treatment he will have received.

• Evaluations and measurements:

Patients will be required to perform functional tests of the upper limb (Wolf Motor Function Test (WMFT)), filmed and timed, a test of spasticity (Tardieu) as well as to answer certain questionnaires concerning their perception of the evolution of the disease and their disability (Stroke Impact Scale, Barthel Index), their emotional state (HADS), if they have experienced side effects, sensitivity test with monofilaments or Semmes and Weinstein test, the Fugl Meyer, the timed up and go, the test of 10m, the four step square test, the berg balance scale, the postural assessment scale and the trunk impairment scale. These evaluations will take place at Day 0 (corresponding to the first day after the 48h of strict bedtime), Day 7, 15, 30, 90, 6 months and 1 year. They will be done in two stages, on two successive days, so as not to exhaust the patient.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man
* Between 18 and 80 years old
* First ever stroke
* Capable of signing the consent form

Exclusion Criteria:

* One on the TSST (in high and relatively high risk sections)
* Previous neurological or orthopedic pathologies affecting limbs
* Cognitive deficits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test Change | 48 hours post onset, 7, 14, 21 and 28 days post onset, 3 and 6 months post onset and 1 year post onset
  Functional outcome of the paretic limb
Semmes Weinstein Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Monofilament sensory test
Timed up and go Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  walking test
10 meter walk test Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Walking speed test

SECONDARY OUTCOMES:
Tardieu spasticity scale Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  spasticity scale, the higher the score the higher the spasticity
Stroke impact scale Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Scale measuring impact of stroke on life, the higher the score the higher the worse off the patient is
HADS Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Depression and anxiety scale, the higher the score the higher the more depressed or anxious the patient is
Fugl Meyer Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Upper and lower limb motor outcomes, the higher the score the higher the better the patient is
4 square step test Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Balance test, the higher the score the higher the worse the patient is
Berg Balance scale Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Balance test, the higher the score the higher the score, the better the patient is
Postural assessement scale Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  Balance test, the higher the score the higher the better the patient is
Trunk impairment scale Change | 48 hours post onset, days 7, 14, 21 and 28 post onset, 3 and 6 months post onset and 1 year post onset
  balance test, the higher the score the higher the better the patient is

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bornheim, Msc, Principal Investigator — Liege Univeristy Hospital
Locations (1):
- Liege Univeristy Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No